CLINICAL TRIAL: NCT05541939
Title: Phase 2 Randomized Single Ascending Dose Study in Post-Bariatric Hypoglycemia Subjects to Determine the Effect of Mizagliflozin Formulations on Postprandial Glucose and Insulin Levels
Brief Title: Effect of Mizagliflozin on Postprandial Glucose and Insulin in Post-Bariatric Hypoglycemia Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vogenx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VGX-001-011
Record Dates: First submitted 2022-09-08; First posted 2022-09-15 (Actual); Results first posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-05

CONDITIONS: Postbariatric Hypoglycemia
MeSH Terms: interventions — mizagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm A (Experimental): Subjects will receive two separate single doses (Period 1 and Period 2) of encapsulated mizagliflozin
  Interventions: Drug: Mizagliflozin
- Treatment Arm B (Experimental): Subjects will receive one dose of liquid formulation (Period 1), and one dose (optional) of encapsulated mizagliflozin (Period 2)
  Interventions: Drug: Mizagliflozin

INTERVENTIONS:
Drug: Mizagliflozin — Encapsulated or Liquid Formulation

SUMMARY:
This clinical study will examine the safety and tolerability, as well as the effects of orally administered mizagliflozin on post prandial glucose and insulin levels in subjects diagnosed with post-bariatric hypoglycemia (PBH).

DETAILED DESCRIPTION:
This is a Phase 2 randomized, sequential crossover single ascending dose study in PBH subjects to determine the effect of two mizagliflozin formulations This study will examine single doses of mizagliflozin in either a liquid or encapsulated formulation. Subjects will be randomly assigned to one of two treatment arms. Safety, tolerability and pharmacodynamic response to mizagliflozin will be assessed in subjects during a mixed meal tolerance test (MMTT).

ELIGIBILITY:
Inclusion Criteria:

* Roux-en-Y gastric bypass surgery performed > 6 months prior to enrollment
* Diagnosis of PBH

Exclusion Criteria:

* History of current medical conditions (other than PBH) which may result in hypoglycemia such as insulinoma, adrenal insufficiency, insulin autoimmune hypoglycemia, congenital hyperinsulinemia.
* Current use of insulin or insulin secretagogues.
* History of current dumping syndrome.
* History of current fasting hypoglycemia.
* Pregnancy and/ or Lactation: For women of childbearing potential: there is a requirement for a negative urine pregnancy test and for agreement to use contraception during the study and for at least 2 weeks after participating in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Stanford, Palo Alto, California
  - University of Colorado / Anschutz Medical Campus, Aurora, Colorado

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 9 participants were screened between September 2022 and January 2023. 7 participants at University of Colorado/Anschutz Medical Campus and 2 participants at Stanford.University
Pre-assignment Details: All 9 screened participants met eligibility criteria and were randomized
Groups:
- Treatment Arm A: Randomized participants received a Baseline MMTT. After approximately 7 days the participants returned to the clinic for Period 1 treatment, a single 2.5 mg capsule of mizagliflozin, followed by an MMTT. After a 7-day washout, participants returned to the clinic for Period 2 treatment, a single 5.0 mg capsule of mizagliflozin, followed by an MMTT.
- Treatment Arm B: Randomized participants received a Baseline MMTT. After approximately 7 days the participants returned to the clinic for Period 1 treatment, a single 2.5 mg liquid formulation of mizagliflozin, followed by an MMTT. After a 7-day washout, participants returned to the clinic for Period 2 treatment, a single 10.0 mg capsule of mizagliflozin, followed by an MMTT.
Period: Overall Study
Arm/Group | Treatment Arm A | Treatment Arm B
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Arm A: Randomized participants received a Baseline MMTT. After approximately 7 days the participants returned to the clinic for Period 1 treatment, a single 2.5 mg capsule of mizagliflozin, followed by an MMTT. After a 7-day washout, participants returned to the clinic for Period 2 treatment, a single 5.0 mg capsule of mizagliflozin, followed by an MMTT.
  Mizagliflozin: Encapsulated
- Total: Total of all reporting groups
Arm/Group | Treatment Arm A | Treatment Arm B | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 4 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 4 | 3 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Baseline MMTT (pharmacodynamic assessment for glucose and insulin) [Count of Participants; unit: Participants] | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Glucose Nadir After Mizagliflozin Dosing
Description: Time course of glucose concentrations during MMTT
Time Frame: 0-3 hours following liquid meal
Population: Change from Baseline MMTT in Glucose Nadir (mg/dL)
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Treatment Arm A: Subjects will receive two separate single doses (Period 1 and Period 2) of encapsulated mizagliflozin
  Mizagliflozin: Encapsulated
- Treatment Arm B: Subjects will receive a single dose of liquid formulation (Period 1) and a single dose of encapsulated (Period 2)
Arm/Group | Treatment Arm A | Treatment Arm B
Number analyzed (Participants) | 5 | 4
mg/dL
  2.5 mg Capsule: number analyzed (Participants) | 5 | 0
  2.5 mg Capsule | 6.2 (14.8) |
  5.0 mg Capsule: number analyzed (Participants) | 5 | 0
  5.0 mg Capsule | 4.0 (17.7) |
  2.5 mg Liquid: number analyzed (Participants) | 0 | 4
  2.5 mg Liquid |  | 17.5 (30.5)
  10.0 mg Capsule: number analyzed (Participants) | 0 | 4
  10.0 mg Capsule |  | 31.5 (29.0)

ADVERSE EVENTS:
Time Frame: 34 Days
Groups:
- Treatment Arm A Period 1 (2.5 mg Capsule): Subjects will receive a single 2.5 mg capsule
  Mizagliflozin: Encapsulated
- Treatment Arm A Period 2 (5.0 mg Capsule): Subjects will receive a single 5.0 mg capsule
  Mizagliflozin: Encapsulated
- Treatment Arm B Period 1 (2.5 mg Liquid Formulation): Subjects will receive a single 2.5 mg liquid formulation
  Mizagliflozin: Liquid Formulation
- Treatment Arm B Period 2 (10.0 mg Capsule): Subjects will receive a single 10.0 mg capsule
  Mizagliflozin: Encapsulated
Arm/Group | Treatment Arm A Period 1 (2.5 mg Capsule) | Treatment Arm A Period 2 (5.0 mg Capsule) | Treatment Arm B Period 1 (2.5 mg Liquid Formulation) | Treatment Arm B Period 2 (10.0 mg Capsule)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 4/5 | 1/5 | 2/4 | 2/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm A Period 1 (2.5 mg Capsule) (N=5) | Treatment Arm A Period 2 (5.0 mg Capsule) (N=5) | Treatment Arm B Period 1 (2.5 mg Liquid Formulation) (N=4) | Treatment Arm B Period 2 (10.0 mg Capsule) (N=4)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hunger (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lack of satiety (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Taste disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT05541939/Prot_SAP_000.pdf